CLINICAL TRIAL: NCT05336539
Title: A Community Population Screening Cohort Study Based on Polygene Methylation Detection for Colorectal Cancer in Yangzhou
Status: Recruiting | Type: Observational
Sponsor: Singlera Genomics Inc. (Industry)
Collaborators: Northern Jiangsu People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PreC
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer
Keywords: Polygenic methylation; The community crowd; Colorectal cancer screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Positive group: subjects received colorectal cancer polygene methylation test at baseline, and all positive results were included in the positive group. They will undergo further FIT testing, blood carcinoembryonic antigen testing and colonoscopy within three months of colorectal cancer polymethylation testing.

SUMMARY:
This is a cross-sectional cohort study based on community population jointly developed by Northern Jiangsu People's Hospital and Shanghai Kunyuan Biological Technology Co., LTD. This study will verify the real world results of polygene methylation detection of colorectal cancer in a large prospective cohort of community population, which is expected to enroll 80,000 permanent residents in Yangzhou city. The preliminary design period of the study is 5 years. In this study, questionnaire survey and polygene methylation test of colorectal cancer were used as the primary screening method, and colonoscopy was used as the further validation examination method to screen colorectal cancer and precancerous lesions. The diagnosis and outcome of all lesions were based on colonoscopy and pathological examination. The evaluation indexes include sensitivity, specificity, detection rate of precancerous lesions and adenoma.

DETAILED DESCRIPTION:
The study is expected to complete baseline examinations of 80,000 subjects within 1 year. Community members who sign informed consent forms will complete the Colorectal cancer Risk Factor Assessment Questionnaire, history collection, and colorectal cancer polymethylation test early screening at baseline. Subjects who tested positive for polygene methylation screening for colorectal cancer will undergo a fecal immunochemistry (FIT) test, a blood carcinoembryo antigen (CEA) test, and colonoscopy within 3 months. Telephone follow-up medical history was collected at 1, 2, 3, and 4 years after baseline, and telephone follow-up survival outcomes were studied at 5 years after baseline. During the follow-up, patients diagnosed with colorectal cancer by colonoscopy will reach the study end point, and patients treated with polyps or adenomas found during colonoscopy will also reach the study end point.

ELIGIBILITY:
Inclusion Criteria:

* 1) Permanent resident population of Yangzhou; 2) Chronological age: 40~74 years, including critical value (refer to birth date of id card); 3) Have full capacity of conduct; 4) After enrollment, they could voluntarily cooperate to complete the Colorectal cancer Risk Factor Assessment Questionnaire and accept telephone follow-up; 5) Agree to timely feed back the information related to tumor diagnosis to the investigator during the study process; 6) Willing and able to sign informed consent.

Exclusion Criteria:

* 1) History of colorectal cancer and other malignant tumors; 2) previous colorectal resection; 3) are receiving any cancer-related treatment; 4) Those who have received major surgical treatment such as blood transfusion and transplantation within 3 months; 5) Participate in other interventional clinical investigators within 3 months; 6) Pregnant or lactating women; 7) Patients with autoimmune diseases, genetic diseases, mental diseases/disabilities and other diseases considered unsuitable for the study by the researcher; 8) Poor compliance, unable to complete the study according to the judgment of the researcher.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects of this study were permanent residents in Yangzhou who met the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 80000 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of polygenic methylation detection in colorectal cancer | assessed up to 5 years
  To evaluate the sensitivity, specificity, and positive/negative predictive value of polygenic methylation tests for colorectal cancer in subjects
Application value of polygene methylation detection in colorectal cancer in community population | assessed up to 5 years
  To verify the effectiveness and clinical value of this detection method in the diagnosis of colorectal cancer in yangzhou community population.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Jun, Master, Study Director — Northern Jiangsu People's Hospital，Yangzhou，China; Liu Rui, Doctor, Principal Investigator — Singlera Genomics Inc.
Locations (2):
- China (2):
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Yangzhou First People's Hospital, Yangzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo S, Diep D, Plongthongkum N, Fung HL, Zhang K, Zhang K. Identification of methylation haplotype blocks aids in deconvolution of heterogeneous tissue samples and tumor tissue-of-origin mapping from plasma DNA. Nat Genet. 2017 Apr;49(4):635-642. doi: 10.1038/ng.3805. Epub 2017 Mar 6. PMID 28263317
- [Derived] Wang B, Zhang Y, Liu J, Deng B, Li Q, Liu H, Sui Y, Wang N, Xiao Q, Liu W, Chen Y, Li Y, Jia H, Yuan Q, Wang C, Pan W, Li F, Yang H, Wang Y, Ding Y, Xu D, Liu R, Fang JY, Wu J. Colorectal cancer screening using a multi-locus blood-based assay targeting circulating tumor DNA methylation: a cross-sectional study in an average-risk population. BMC Med. 2024 Nov 27;22(1):560. doi: 10.1186/s12916-024-03777-2. PMID 39604913